CLINICAL TRIAL: NCT02368067
Title: Study of Instillation Technique Using The Modified Intra- Uterine Manipulator Catheter With Methylene Blue, Isosulfan Blue or Indocyanine Green Dyes, Compared to Cervical Injection, For Sentinel Lymph Node Detection in Endometrial Carcinoma
Brief Title: Improved Method of Detecting Cancer Metastases
Acronym: SITs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Southeastern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SERMC- Endometrial Carcinoma
Record Dates: First submitted 2014-11-17; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care Sentinal Node Dye (Active Comparator): Surgery route, as determined by the patient and clinician, will determine which standard clinical dye will be used.
  Interventions: Procedure: Standard of Care Sentinal Node Dye
- Installation of Study Sentinal Node Dye (Experimental): Surgery route, as determined by the patient and clinician, will determine which study dye will be used for delivery by the experimental route.
  Interventions: Procedure: Study Sentinal Node Dye

INTERVENTIONS:
Procedure: Standard of Care Sentinal Node Dye — Delivery of sentinal node dye by different routes
  Arms: Standard of Care Sentinal Node Dye
Procedure: Study Sentinal Node Dye — Patients will receive different types of dye by different routes of administration
  Arms: Installation of Study Sentinal Node Dye

SUMMARY:
The purpose of this study is to compare the Instillation Technique Using The Modified Intra- Uterine Manipulator Catheter With Methylene Blue, Isosulfan Blue or Indocyanine Green Dyes, Compared to Cervical Injection, For Sentinel Lymph Node Detection in Endometrial Carcinoma.

DETAILED DESCRIPTION:
Following consent, surgery will be determined by the physician thereby determining group assignment- i.e the laparoscopic surgery group oror the robotic assisted surgery group. Both groups will undergo SLN mapping by instillation and injection. The Laparotomy/Laparoscopy Group will have Lymphazurin by injection and instillation of methylene blue dye. The Robot Assisted Group will have ICG by injection and instillation of methylene blue. Patients will undergo total hysterectomy, bilateral salpingoophorectomy, pelvic and paraaortic lymphadenectomy through laparotomy, laparoscopic or robotic assisted surgery as clinically determined by their attending physician. Subjects will undergo this surgery whether or not enrolled in the study.

Any clinically indicated uterine manipulator will be acceptable. Potential subjects will be informed of the potential risks of this device so they may make an informed decision about participation in the study. However the manipulator is standard of care and is not a study related risk. Subjects who agree to this study procedure will be monitored for adverse events.

The dyes used in this study are commercially available and will be provided through internal funding from the CTCA Gynecology/Oncology Department. Potential subjects will be informed

of the potential risks of these drugs so they may make an informed decision about participation in the study. Subjects who agree to this study procedure will be monitored for adverse events.

After administration of anesthesia, the intra-uterine uterine manipulator catheter will be inserted using the following suggested instructions for use;

• After the standard of care vaginal prep with povidone-iodine or any other surgeon preference cleansing solution, expose the cervix using a vaginal speculum. No additional preparation of the cervix is needed.

Immediately following exposure pf the cervix with the speculum, and before introduction of the intra-uterine uterine manipulator with catheter, 4ml total of isosulfan 1% blue or ICG (depending on what route of surgery is being elected) dye will be delivered by cervical injection as follows:

* Using a 20 or 22 gauge spinal needle, inject dye into the cervix at the 12, 3, 6 and 9 o'clock positions.
* Each site will receive approximately 1ml of dye with ½ superficial just under the mucosa and the remainder approximately 1cm deep to the prior injection.

The 22 gauge needles are commercially available and will be provided as routine clinical care. Potential subjects will be informed of the potential risks of injection so they may make an informed decision about participation in the study. Subjects who agree to this study procedure will be monitored for adverse events.

• Introduce the uterine manipulator with catheter trans-cervically until the distal balloon is positioned in the lower portion of the uterus. This is no different from routine clinical care.

Immediately following cervical injection and placement of the uterine manipulator and once intra-abdominal, the first step in surgery will be to occlude both fallopian tubes, as typically done as part of this surgery, using electrocautery devices (e.g. Ligasure) for sealing only the tubes.

Immediately following occlusion of both fallopian tubes, the comparator instillation dye will be instilled into the uterine cavity through the pre-inserted intra-uterine uterine manipulator catheter as follows:

* Insert the clinically selected uterine manipulator as per standard clinical practice.
* Slowly inject the dye through the center uterine cavity catheter access port., Rapid injection of dye could cause high intrauterine pressure resulting in extravasation. Use slow constant pressure to instill the dye. This can be done by the surgical assistant or by the operating surgeon via a long extension tubing.

It is estimated that it may take up to 40 minutes for the dyes to be absorbed by the surrounding tissue and taken up by the lymphatic vessels turning the nodes blue or green. During this time

the surgery will proceed without delay. These study procedures will not increase the estimated total time to perform the surgery.

The surgery will proceed as routine for any sentinel node dissection. Briefly, during regular dissection, visual identification of any dye taken up by any nodes and specific anatomical distributions will be documented using an anatomical documentation sheet.

Visual detection of the methylene and isosulfan blue dye will be done with the investigator's naked eye.

Visual detection of ICG dye will include use of a charge-coupled device (CCD) camera called Spycam equipped with 3 main components (a near-infrared sensitive image intensifier, 16-bit dynamic-range frame transfer CCD camera and light-emitting diodes [LEDs] that is mounted to the robotic surgical instruments. The Spycam will be directed onto the operative field illuminating the fluorescing dye green. The camera is connected to a monitor and images will display on the screen and will be analyzed using digital imaging processing.

Using the clock in the surgery room as a reference, a member of the surgical team will record the exact time elapsed (in minutes) from administration until visual detection of dye is made for each technique. Blue/green nodes will be labeled as sentinel nodes and non-blue/green nodes will be labeled as non-sentinel. Blue/green nodes will also be labeled to describe which dye is being detected (methylene, isosulfan or ICG). Differences in the dye deposition/absorption by each method (injection vs. instillation) will be documented as either detected or not detected in the nodes and channels using color photography in the surgical setting. Continuous monitoring will be done for adverse events during the surgery and post operatively up to time of patient discharge from the hospital.

All node samples will be histopathologically examined with Hematoxylin and Eosin (H&E) and Immunohistochemistry (IHC) staining to detect micro-metastasis. Analysis will compare results of the instillation technique to cervical injection technique in the same subject for sensitivity of SLN mapping, estimating the false negative predictive value, time to detect SLNs, anatomical distributions of the SLNs, and differences in dye absorption using each technique.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old at the time of consent.
* Preoperatively diagnosed endometrial carcinoma of any stage or grade and planned to undergo surgery (laparotomy, laparoscopy or robotic assisted) at IUSCC.
* Medically operable status.
* Ability to understand and willingness to sign a written informed consent and authorization for the release of health information.

Exclusion Criteria:

* Previous radiotherapy.
* Previous retroperitoneal surgery.
* Significant physical limitations preventing proper vaginal examination as determined by the treating physician.
* Personal history of allergy to iodides, iodine or shellfish.
* No clinical indication for intra-uterine manipulator use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of sentinel nodes detected by each method. | 1 Year
  To determine if the new procedure is better than the current method of sentinal node detection. We will determine which dye and which route is most sensitive for detected metastatic cancer. Each Sentinel node dye and route will be compared to the full node dissection result.

SECONDARY OUTCOMES:
Time to detection of 1st SN by each method. | 1 year
Sensitivity of each method compared to full node dissection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Del Priore, MD, Principal Investigator — Southeastern Regional Medical Center
Locations (1):
- Southeastern Regional Medical Center, Newnan, Georgia, United States